CLINICAL TRIAL: NCT01641705
Title: Analysis of Respiratory Mechanics in Patients With Rheumatoid Arthritis: Effect of Duration of Disease
Brief Title: Analysis of Respiratory Mechanics in Patients With Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitario Pedro Ernesto (Other)
Responsible Party: Principal Investigator, Alvaro Camilo Dias Faria, Professor, Hospital Universitario Pedro Ernesto
Other Study IDs: AR-01
Record Dates: First submitted 2012-03-13; First posted 2012-07-17 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; respiratory mechanics; time of disease
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Control Group: Group of nonsmokers individuals without respiratory disease.
- RA patients 1: RA patients nonsmokers with up to five years of disease.
- RA group 2: RA patients nonsmokers with six to ten years of disease.
- RA group 3: RA patients nonsmokers with eleven to fifteen years of disease.
- RA group 4: RA patients nonsmokers with sixteen or more years of disease

SUMMARY:
Rheumatoid arthritis (RA) is an autoimmune disease of unknown etiology characterized by peripheral polyarthritis, symmetric, which leads to joint destruction and deformity. It is estimated that the RA reaches about 0.5% of the population. According to data from DATASUS, was responsible for 26,671 hospitalizations, 229 deaths and cost exceeding R$ 20 million in 2005-2007.

The main bodily changes are related to joint problems, however, systemic manifestations are also found in organs such as lung and heart. Although cardiovascular diseases are the most responsible of the deaths AR, pulmonary complications are common and account for 10% to 15% of all mortality. Anaya and colleagues point out that the pulmonary involvement contributes significant morbidity and mortality in these patients. Although pulmonary involvement is a frequent manifestation in RA, the prevalence and nature of rheumatoid lung disease has not yet been precisely established. Several lung disorders such as interstitial pulmonary fibrosis, pulmonary nodules and bronchiolitis may ocorrer1. Laitinen et al point out that studies of lung function appear to be a valuable helper for radiography in the evaluation of pulmonary involvement in connective tissue diseases. Previous studies indicate that patients with RA have an increased incidence of abnormal lung function, according to assessments including spirometry, lung volume tests and diffusion capacity of carbon monoxide.

Thus, the main objective of this study is to analyze the respiratory mechanics of patients with RA. Specific objectives were to seek to understand whether a relationship exists between duration of rheumatoid disease and lung function in these patients.

For this, the investigators used 18 subjects in the control group, free of pulmonary disease and / or heart, all nonsmokers. In the RA group, a total of 72 patients divided into 4 groups of 18 volunteers each, classified according to disease duration (0-5 years, 6-10 years, 11-15 years and> or = 16 years). It is noteworthy that all patients in the RA group will also be non-smokers, since it is already known in the literature that smoking impairs lung function. All individuals will perform the function test with a trained technician and qualified to function. The examinations will be conducted: Forced oscillation technique and spirometry, in that order.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers with Rheumatoid Arthritis for Patients Group;
* Volunteers without any respiratory disease for the control group.

Exclusion Criteria:

Smokers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The control group will consist of healthy subjects, nonsmokers, who had no episode of respiratory infection thirty days before the examinations.
  The group of patients with rheumatoid arthritis will be comprised of individuals treated at the Department of Rheumatology (Hospital Universitártio Pedro Ernesto) nonsmokers, who had no episode of respiratory infection thirty days before the examinations.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-12 (Estimated); Study Completion 2013-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro L de Melo, Study Director — State University of Rio de Janeiro
Locations (1):
- Laboratório de Instrumentação Biomédica, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Result] Faria AD, Lopes AJ, Jansen JM, Pinheiro GC, Melo PL. Diagnostic performance of the Forced Oscillation Technique in the detection of early respiratory changes in rheumatoid arthritis. Annu Int Conf IEEE Eng Med Biol Soc. 2010;2010:6034-7. doi: 10.1109/IEMBS.2010.5627605. PMID 21097117
- [Derived] Faria AC, Barbosa WR, Lopes AJ, Pinheiro Gda R, Melo PL. Contrasting diagnosis performance of forced oscillation and spirometry in patients with rheumatoid arthritis and respiratory symptoms. Clinics (Sao Paulo). 2012 Sep;67(9):987-94. doi: 10.6061/clinics/2012(09)01. PMID 23018292